CLINICAL TRIAL: NCT03717402
Title: Smartphone Technology to Alleviate Malignant Pain (STAMP): Development and Piloting of a Novel mHealth Intervention to Support Cancer Patients, Nurses, and Physicians in Opioid Management
Brief Title: Smartphone Technology to Alleviate Malignant Pain (STAMP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Andrea Enzinger, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-504; 1R21NR017745-01 (NIH)
Record Dates: First submitted 2018-10-18; First posted 2018-10-24 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Cancer; Pain Management; Opioid Use
Keywords: Cancer; Pain management; Opioid use; Health app; Gastrointestinal cancer; Breast cancer; Lung cancer
MeSH Terms: conditions — Neoplasms; Agnosia; Gastrointestinal Neoplasms; Breast Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Participants (Other): Patients with advances cancer using opioids for chronic pain will be enrolled and asked to use the STAMP cancer pain management app for 4 weeks.
  Interventions: Behavioral: Intervention Participants

INTERVENTIONS:
Behavioral: Intervention Participants — Patients with advances cancer using opioids for chronic pain will be enrolled and asked to use the STAMP cancer pain management app for 4 weeks.

SUMMARY:
The purpose of the study is to develop the STAMP app (Smartphone Technology to Alleviate Malignant Pain). This app will be used by patients with advanced cancer to track symptoms and receive tailored symptom management advice.

This is a single arm pilot feasibility study of the application among patients with advanced cancer and chronic pain who are using opioids in the home setting. Patients will be asked to use the application for a four week period. Clinicians responsible for the patients' pain management will be asked to review alerts from the STAMP system and respond accordingly. The primary outcomes of the study relate to feasibility and acceptability.

DETAILED DESCRIPTION:
A pilot study will be conducted at DFCI to demonstrate the utilization and efficacy of the STAMP app among patients with chronic cancer pain and their cancer care providers. This will be a single arm study with up to 20 patients. Patients with advanced solid tumors who are using opioids to manage chronic cancer pain will be recruited from outpatient clinics (palliative care), and they will be asked to use the app for 4 weeks. Once a patient is enrolled in the study, a research assistant (RA) will set up the app, putting in the patient's prescribed opioids and laxatives. Patient will have access to educational materials about pain management and patient educational videos about pain management and opioids through the app. Patient will be prompted to take daily surveys for symptom reporting and medication updates. At the end of each survey patients receive, a summary of their symptom severity, with links to tailored educational content about pain management, and recommendations about how to safely titrate over-the-counter laxatives to manage opioid-induced constipation. This laxative advice operates within the parameters of normative and approved over-the-counter laxative use, and has been extensively reviewed, vetted, and approved by multidisciplinary groups of clinicians. If patients report any severe symptoms, they are instructed to contact their care team immediately, with a telephone number included on the application screen. If patients' pain is poorly controlled but not severe enough to be prompted to immediately contact their care team (for example if their average pain is above a 4 and not acceptable), they are reminded to contact their care teams if their symptoms worsen or they are concerned about it. Finally, if they report any concerning abdominal symptoms (e.g. no bowel movement in 4 or more days, haven't passed gas from bottom or ostomy, new or severe abdominal pain, vomiting two or more times in the past 24 hours), patients are not given any laxative titration instructions and are instead advised to contact their care team for more advice.

The research team will monitor the portal where patient survey responses are presented. If a severe symptom is reported, the research team will contact the relevant nursing staff for clinical follow-up (as per the above paragraph, patients are always advised to contact their care teams for safety concerns, and there is no expectation for immediate nurse outreach). Nurses and physicians involved in the care of participating patients will also have access to patient-responses on the clinician portal.

Participants will complete a brief survey at baseline and again at end of study (4 weeks). They will also be offered an optional qualitative debriefing at end of study.

ELIGIBILITY:
Inclusion Criteria:

Patient Inclusion Criteria:

* Patient is cared for within participating clinic (PC)
* Age ≥21
* Diagnosed with locally advanced, metastatic solid tumor, or multiple myeloma being managed with palliative intent
* Chronic pain related to cancer or cancer treatment, persisting or at least two weeks
* Average pain rating of ≥4/10 currently, or at least one day within the past week
* Active prescription for short and/or long acting opioids
* Takes at least 1 opioid medication on most days
* Own a compatible smartphone:
* iPhone, have updated or willing to update it to the past 3 iOS version releases
* Android flagship devices with more than 5% market share, last 2 android version releases

Clinician Inclusion Criteria:

* Physicians and mid-level providers practicing in participating clinics and caring for a patient on the study
* Nurse Navigators working within participating clinics

Exclusion Criteria:

Patient Exclusion Criteria:

* Cognitive impairment that would interfere with study participation, as judged by treating clinician
* Inability to speak English
* History of opioid use disorders
* Enrolled in hospice
* Currently hospitalized
* Use of opioids not supported by STAMP
* Pain primarily related to a recent surgery
* Currently has or has had recurrent bowel obstructions
* The following special populations are excluded: adults unable to consent, prisoners, and pregnant women.

Clinician Exclusion Criteria:

- Unwilling to participate

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Enzinger, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van den Beuken-van Everdingen MH, Hochstenbach LM, Joosten EA, Tjan-Heijnen VC, Janssen DJ. Update on Prevalence of Pain in Patients With Cancer: Systematic Review and Meta-Analysis. J Pain Symptom Manage. 2016 Jun;51(6):1070-1090.e9. doi: 10.1016/j.jpainsymman.2015.12.340. Epub 2016 Apr 23. PMID 27112310
- [Background] Dalal S, Bruera E. Access to opioid analgesics and pain relief for patients with cancer. Nat Rev Clin Oncol. 2013 Feb;10(2):108-16. doi: 10.1038/nrclinonc.2012.237. Epub 2013 Jan 15. PMID 23319138
- [Background] Jadad AR, Browman GP. The WHO analgesic ladder for cancer pain management. Stepping up the quality of its evaluation. JAMA. 1995 Dec 20;274(23):1870-3. PMID 7500538
- [Background] Deandrea S, Montanari M, Moja L, Apolone G. Prevalence of undertreatment in cancer pain. A review of published literature. Ann Oncol. 2008 Dec;19(12):1985-91. doi: 10.1093/annonc/mdn419. Epub 2008 Jul 15. PMID 18632721
- [Background] Breivik H, Cherny N, Collett B, de Conno F, Filbet M, Foubert AJ, Cohen R, Dow L. Cancer-related pain: a pan-European survey of prevalence, treatment, and patient attitudes. Ann Oncol. 2009 Aug;20(8):1420-33. doi: 10.1093/annonc/mdp001. Epub 2009 Feb 24. PMID 19244085
- [Background] Cleeland CS, Gonin R, Hatfield AK, Edmonson JH, Blum RH, Stewart JA, Pandya KJ. Pain and its treatment in outpatients with metastatic cancer. N Engl J Med. 1994 Mar 3;330(9):592-6. doi: 10.1056/NEJM199403033300902. PMID 7508092
- [Background] Tariman JD, Berry DL, Halpenny B, Wolpin S, Schepp K. Validation and testing of the Acceptability E-scale for web-based patient-reported outcomes in cancer care. Appl Nurs Res. 2011 Feb;24(1):53-8. doi: 10.1016/j.apnr.2009.04.003. Epub 2009 Sep 18. PMID 20974066
- [Derived] Azizoddin DR, Hassett M, Anderson KS, Kessler D, Wright A, Gorra M, Kematick B, Chua I, Brandoff D, Lally K, Nabati L, MacIsaac S, Tulsky JA, Enzinger A. MyPainPal, a Novel mHealth App to Improve Pain in Patients With Advanced Cancer: Single-Arm Pilot Study. JMIR Cancer. 2025 Dec 30;11:e79942. doi: 10.2196/79942. PMID 41468579

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 20 participants where consented and enrolled on this single-arm intervention study.
Groups:
- Intervention Participants: Patients with advanced cancer using opioids for chronic pain will be enrolled and asked to use the STAMP cancer pain management app for 4 weeks.
Period: Overall Study
Arm/Group | Intervention Participants
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0
  Asian | 2
  Black or African American | 2
  Native Hawaiian or Other Pacific Islander | 0
  White | 16
  I don't know | 0
Ethnicity [Count of Participants; unit: Participants]
  Non-Hispanic/LatinX | 20
  Hispanic/LatinX | 0
Education [Count of Participants; unit: Participants]
  Some high school | 0
  High school diploma | 3
  Some college (AA, other) | 6
  College degree (BA, BS, other) | 5
  Higher level degree (MA, MS, MD, PhD, other) | 5
  Missing | 1
Marital Status [Count of Participants; unit: Participants]
  Single | 1
  Married | 17
  Widowed | 0
  Separated | 1
  Divorced | 1

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Patient Log Ins
Description: We will calculate the frequency that patients log in to the application using simple descriptive statistics.
Time Frame: 4 Weeks
Measure: Median (Inter-Quartile Range); unit: log ins to the application per patient
Arm/Group | Intervention Participants
Number analyzed (Participants) | 20
log ins to the application per patient | 14 [9 to 17]

2. Primary Outcome: Frequency of Symptom Survey Completion
Description: We will calculate the number of times patients completed a symptom survey on app during their 28 days on study. Patients could complete up to one symptom survey per day on study.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: completed symptom survey(s) per patient
Arm/Group | Intervention Participants
Number analyzed (Participants) | 20
completed symptom survey(s) per patient | 8 [5 to 14]

3. Secondary Outcome: E-scale Acceptability
Description: Patients will rate overall acceptability of the application using a modified acceptability e-scale. This 6-item measure asks patients to rate the app on ease of use, understandability, enjoyment, helpfulness, time spent, and overall satisfaction, on a 1 to 5 Likert scale. Items are summed to for a total score, ranging from 6 to 30 with 30 being the highest acceptability score.
Time Frame: 4 Weeks
Measure: Mean (Standard Deviation); unit: score on the acceptability scale
Arm/Group | Intervention Participants
Number analyzed (Participants) | 20
score on the acceptability scale | 24 (4.37)

4. Secondary Outcome: Usability
Description: Patients will complete a validated 10-item system usability scale (SUS) with total scores ranging from 0-100, where a score of 100 being the best possible usability score.
Time Frame: 4 Weeks
Measure: Mean (Standard Deviation); unit: score on the SUS scale
Arm/Group | Intervention Participants
Number analyzed (Participants) | 20
score on the SUS scale | 78.3 (16.2)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention Participants
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Participants (N=20)
Consent form error (Social circumstances) | 20 (20) — An outdated version of the informed consent document was used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/02/NCT03717402/Prot_SAP_000.pdf